CLINICAL TRIAL: NCT02011139
Title: Effectiveness of Cognitive-behavioral Group Therapy for Enhancing Mental Health and Quality of Life in Maintenance Hemodialysis Patients
Brief Title: Cognitive-behavioral (CBT) in ESRD Patients With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Boramae Hospital (Other)
Responsible Party: Principal Investigator, Chun Soo Lim, Professor, Seoul National University Boramae Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CBT-ESRD
Record Dates: First submitted 2013-12-03; First posted 2013-12-13 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Kidney Failure, Chronic; Depression; Quality of Life
MeSH Terms: conditions — Kidney Failure, Chronic; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): 12 sessions of Cognitive-behavioral group therapy in the first 12 weeks
  Interventions: Behavioral: Cognitive-behavioral group therapy
- Group B (Active Comparator): 12 sessions of Cognitive-behavioral group therapy in the second 12 weeks
  Interventions: Behavioral: Cognitive-behavioral group therapy

INTERVENTIONS:
Behavioral: Cognitive-behavioral group therapy

SUMMARY:
Depression is common in end-stage renal disease (ESRD) patients and has a negative effect on the quality of life, functional ability, and mortality, with a prevalence rate as high as 20-25%. However, it is hard to use anti-depressant due to the safety issue, and there has been little data so far particularly in terms of randomized clinical trials. Here, we investigate the effect of cognitive-behavioral group therapy for enhancing mental health and quality of life in patients with ESRD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage renal disease : on hemodialysis more than 3 months
* Patients with BDI-II score >= 15 points
* Adult with age >= 20 years old
* Patients who were able to understand and willing to sign the written informed consent

Exclusion Criteria:

* Patients on hemodialysis due to acute kidney injury
* Patients who are on admission
* Patients who are undergoing chemotherapy or radiation therapy due to progressive malignant disease
* Patients who are planning kidney transplantation within few months
* Patients with cognitive dysfunction, mental retardation, and drug addict
* Patients who are unavailable for adequate communication with researchers
* Patients who changed anti-depressive agent or dose within 2 months before/after the trial

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) score | 3 months

SECONDARY OUTCOMES:
Secondary assessment tools for depression,anxiety, and quality of life | 3 months
  Hamilton Depression Rating Scale (HAMD-17): assessment for depressive mood
Secondary assessment tools for depression,anxiety, and quality of life | 3 months
  Beck Anxiety Inventory (BAI)
Secondary assessment tools for depression,anxiety, and quality of life | 3 months
  The Perceived Stress Scale
Secondary assessment tools for depression,anxiety, and quality of life | 3 months
  KD-QOL: quality of life related with kidney disease
Secondary assessment tools for depression,anxiety, and quality of life | 3 months
  WHOQOL_BREF: overall quality of life
Secondary assessment tools for depression,anxiety, and quality of life | 3 months
  Temperament and Character Inventory (TCI)
Secondary assessment tools for depression,anxiety, and quality of life | 3 months
  Diagnosis of major depressive disorder by DSM-IV
Secondary assessment tools for depression,anxiety, and quality of life | 3 months
  Biomarker related with depression: serotonin level and etc.
Secondary assessment tools for depression,anxiety, and quality of life | 3 months
  Additional anti-depressant use after trial

CONTACTS AND LOCATIONS:
Overall Officials: Chun Soo Lim, M.D. PhD, Principal Investigator — Seoul National University Boramae Hospital
Locations (1):
- Seoul National University Boramae Hospital, Seoul, South Korea